CLINICAL TRIAL: NCT04589442
Title: A Prospective, Randomized Study to Evaluate the Effectiveness of Microsurfaced vs Control Cadaveric Decellularized Grafts to Establish Wound Bed Preparedness in Deep Partial and Full Thickness Burn Wounds
Brief Title: Microsurfaced Grafts in Deep Burn Wounds
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CellTherX (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MB2019-01
Record Dates: First submitted 2020-10-05; First posted 2020-10-19 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Burns; Wound Heal
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of Care Dermal Graft (Active Comparator): Standard of care cryopreserved cadaveric split thickness skin grafts
  Interventions: Biological: Split thickness skin graft
- Standard of Care Dermal Graft - Microsurfaced (Experimental): Microsurfaced cryopreserved cadaveric split thickness skin grafts
  Interventions: Biological: microsurfaced split thickness skin graft

INTERVENTIONS:
Biological: Split thickness skin graft — standard of care graft
  Arms: Standard of Care Dermal Graft
Biological: microsurfaced split thickness skin graft — standard of care graft that has been microsurfaced
  Arms: Standard of Care Dermal Graft - Microsurfaced

SUMMARY:
This study is designed as a prospective, randomized, within subject controlled design to evaluate the effectiveness of Microsurfaced vs Control cadaveric grafts for coverage of acute deep-partial or full-thickness burn wounds to promote wound healing. This study will be performed in 2 parts: Time to wound bed preparedness through 6 weeks (Part A) and wound site healing, graft take and long-term scar outcomes (Part B). Subjects will be treated with both control and microsurfaced cadaveric grafts on adjacent deep-partial or full-thickness burn wounds.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by patient or Legally Authorized Representative (LAR)
* Subject with deep partial or full thickness burn injury due to flame burn, scald injury or contact burn
* Study burn site large enough to accommodate placement of control and microsurfaced cadaveric graft (minimum 4 cm2 each) at the same location OR 2 study burn sites large enough to each accommodate control and microsurfaced cadaveric graft, respectively at minimum 4 cm2.
* Total Body Surface Area burned (TBSA) total ≤30 %
* Admission within 72 hours of burn injury
* Non-infected wound as diagnosed by the attending physician upon admission
* Treated as an outpatient or in an observational setting
* 21 years of age or older

Exclusion Criteria:

* Burns involving the face
* Causes other than contact burn, flame or scald injuries (i.e., electrical, chemical or frostbite)
* Admission time greater than 72 hours after the injury
* Wounds noted to be infected at admission
* Is pregnant or plans to become pregnant
* Is nursing or actively lactating
* Developmental disability/significant psychological disorder that in the opinion of the investigator could impair the subject's ability to provide informed consent, participate in the study protocol or record study measures, including untreated schizophrenia, bipolar disorder and psychiatric hospitalization within the last 2 years.
* Active alcohol or substance abuse in the opinion of the investigator that could impair the subject's participation in the study protocol or record study materials
* Any medical condition or co-morbidity that in the opinion of the investigator, would prevent successful participation in the study

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-01-04 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Wound bed prep | 6 week
  To compare wound bed preparedness/time to autograft in deep-partial and full thickness burns and burn wound healing in partial thickness burns in burn sites treated with Microsurfaced vs Control cadaveric graft-treated groups through 6 weeks post initial injury.

SECONDARY OUTCOMES:
Infection | Through 12 months
  Incidence of Infection at each treatment study visit
Autograft take | 2 weeks
  Autograft take will be documented as a percentage of the graft by the physician
Tissue oxygenation | 2 weeks
  Tissue oxygenation will be assessed using hyperspectral imaging
Tissue Oxygenation | 6 weeks
  Change in tissue oxygenation at study burn site at the time of autografting as compared to baseline.
Scar assessment | 3, 6, 9, 12 months
  Scar will be assessed using the Patient and Observer Scar Assessment Scale (POSAS)
Tissue oxygenation | 3, 6, 9, 12 months
  Tissue oxygenation will be assessed using hyperspectral imaging

CONTACTS AND LOCATIONS:
Overall Officials: Claus Brandigi, MD, Principal Investigator — Joseph M Still Research Foundation
Locations (1):
- Joseph M Still Research Foundation, Augusta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No